CLINICAL TRIAL: NCT01377948
Title: Phase 1 Study of Anger Control Therapy Augmented With RAGE-Control (Regulate and Gain Emotional-Control)Delivered on an Inpatient Psychiatric Unit
Brief Title: Reducing Aggression in Children and Adolescent on an Inpatient Unit
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gonzalez-Heydrich, Joseph, M.D. (Individual)
Collaborators: Boston Children's Hospital (Other); Harvard University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X10-06-0278
Record Dates: First submitted 2011-06-15; First posted 2011-06-22 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-03

CONDITIONS: Anger; Aggression
Keywords: Anger; Aggression; CBT; Videogame; biofeedback
MeSH Terms: conditions — Aggression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACT with RAGE-Control (Other): all subjects are assigned to this arm. This is an open feasability proof of concept trail with a single experimental group with all subjects receiving the intervention being studied.
  Interventions: Behavioral: ACT with RAGE-Control

INTERVENTIONS:
Behavioral: ACT with RAGE-Control — This is an open trial of ACT with RAGE-Control which is a behavioral intervention. The therapy involves five psychotherapy sessions taking place over five consecutive days.
  Other Names: Cognitive Behavioral Therapy (CBT)

SUMMARY:
The purpose of this study is to determine whether Anger Control Therapy (ACT) with Regulate and Gain Emotional-Control (RAGE-Control) is a feasible behavioral therapy to provide on a pediatric inpatient psychiatric unit.

DETAILED DESCRIPTION:
Aggression and disruptive behavior are the most common reasons for child and adolescent inpatient psychiatric hospitalization. Aggressive children and adolescents who merit admission to inpatient psychiatric hospitals for treatment typically display dramatic problems with self-regulation that interfere with global adaptive functioning. The goal of this study is to teach self-regulation techniques by combining Cognitive Behavioral Therapy with a biofeedback video game in effort to motivate patients to learn and practice these coping skills, which will translate to decreased feelings of anger and aggression while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* consecutive admissions to the psychiatric inpatient unit between the ages of 9 and 17 years of age
* who were not expected to begin or undergo a change >25% to their antipsychotic or mood stabilizing medications
* elevated levels of anger as demonstrated by baseline score on the State Trait Anger Expression Inventory - Child and Adolescent (STAXI-CA) combined State-anger and Trait-anger score greater than 30.

Exclusion Criteria:

* Inability to consent, comprehend, and effectively participate in the study.
* Gross cognitive impairment due to mental retardation, dementia, or intoxication.
* Started on an antipsychotic or mood stabilizing drug within 5 days of beginning the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in State Trait Anger Expression Inventory - Child and Adolescent | change from baseline to just after 5th daily session of the study treatment

SECONDARY OUTCOMES:
Change in Percentage of time playing videogame with heart rate under preset threshold | During videogame play at end of each of the 5 daily sessions of the study treatment
Therapeutic Helpfulness Questionnaire | after session number 5 of the 5 daily study treatment sessions
  To provide information about feasibility, ratings of perceived helpfulness were collected using the Therapeutic Helpfulness Questionnaire5, which elicits both quantitative and qualitative data in three dimensions: 1) the degree to which it is helpful versus hurtful 2) the degree to which the focus of the treatment was helpful 3) overall satisfaction with the treatment. Participants rated each item from 1 = very unhappy or unhelpful to 7 = very happy or helpful.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Wharff, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Sukhodolsky DG, Cardona L, Martin A. Characterizing aggressive and noncompliant behaviors in a children's psychiatric inpatient setting. Child Psychiatry Hum Dev. 2005 Winter;36(2):177-93. doi: 10.1007/s10578-005-3494-0. PMID 16228146